CLINICAL TRIAL: NCT05743751
Title: Prospective Randomized Controlled Study Normothermic Pulse Perfusion Comparing and Hypothermic Machine Perfusion in Margin Deceased Donor Kidney Transplantation
Brief Title: Normothermic Machine Perfusion (NMP) Versus Hypothermic Machine Perfusion (HMP) in Human Kidney Transplantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhang Tianyu (Other)
Responsible Party: Sponsor-Investigator, Zhang Tianyu, Principal Investigator, China-Japan Friendship Hospital
Organization: China-Japan Friendship Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022-NHLHCRF-LX-03
Record Dates: First submitted 2023-01-28; First posted 2023-02-24 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Kidney Transplantation
Keywords: Kidney Transplantation; Normothermic Machine Perfusion; Hypothermic Machine Perfusion

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Participant and care provider were blinded to the interventions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Hypothermic machine perfusion (Active Comparator): After organ acquisition, the donor kidney was trimmed, and then the donor kidney was connected to the cryoperfusion machine (lifeport, which has been used in routine clinical practice in our hospital) for continuous low temperature mechanical perfusion (<8 ℃). The perfusion solution was extracted for proteomic study at 10 min after perfusion and at the end of perfusion.
  Interventions: Device: Hypothermic machine perfusion
- Normothermic machine perfusion (Experimental): After conventional UW perfusion is obtained, the marginal donor kidney is immediately perfused without ischemia at normal temperature. The perfusion time is at least 4 hours (so as to repair the marginal donor kidney). The perfusion solution is as above, and the perfusion solution is loaded into the device authorized in Europe (XVIVO - KidneyAssist ®）， Connect the transplanted renal artery with the device. Take 5ml perfusion solution in advance before perfusion, 5ml perfusion solution every 30min after perfusion, take perfusion solution at the end of perfusion (blood gas analysis for each perfusion solution, and finally perfusion solution for culture), and measure urine volume every hour. After perfusion, the transplanted kidney was disconnected from the perfusion device, and the donor kidney was perfused again with 2L HTK solution, followed by routine transplantation.
  Interventions: Device: Normothermic machine perfusion

INTERVENTIONS:
Device: Normothermic machine perfusion — XVIVO (perfusion company, Gothenburg, Sweden), functions to be included in perfusion equipment, cardiopulmonary bypass machine and neonatal cardiopulmonary bypass machine, including polyethylene pipeline, heating equipment (perfusion temperature 37 ℃), venous pool (venous pressure is 0 mmHg, adjust the height of perfusion pool), centrifugal pump (arterial pressure is set at initial 75 mmHg, maintain 65 mmHg). The perfusion solution contains 215ml of dextran/albumin solution and 400ml of hematocrit, 2ml of 10% calcium gluconate, 1300u/L heparin and 400mg of cefazolin sodium. The oxygen/carbon dioxide ratio is (95%/5%, 2L/min) for continuous perfusion, and pO2 is maintained at 650mmHg during perfusion. During perfusion, continue to use verapamil, amino acid, glucose and insulin. Lactic acid Ringer solution (10ml/h) was used to supplement the lost circulation volume due to urine production during perfusion.
  Arms: Normothermic machine perfusion
Device: Hypothermic machine perfusion — LifePort Kidney Transporter is designed to integrate with the clinical environment by using readily available supplies, requiring minimal user intervention, and by being easy to use. LifePort Kidney Transporter is a portable, isolated kidney perfusion and transport system, designed to support a donated kidney and to maintain the organ in a near-normal physiologic state under hypothermic aseptic conditions. An insulated plastic housing encloses the kidney and perfusate within a LifePort Kidney Transporter Disposable Perfusion Circuit. LifePort Kidney Transporter components include an Ice Container, Pump Deck, Control Panel, Outer Display, Bubble Detectors, External Connections Panel, sensors, and four lithium-ion batteries. Two handles make the unit easy to lift and carry
  Arms: Hypothermic machine perfusion

SUMMARY:
Due to the rising incidence of renal failure and the improvement of organ transplantation technology, the shortage of donor organs has become one of the main problems limiting the development of kidney transplantation. Marginal donor is one of the important ways to extend the donor pool. Normothermic mechanical perfusion (NMP) is a new generation of organ preservation technology, which can maintain the blood supply and at the same time evaluate the marginal kidney function during the organ preservation. However, the clinical effect has not been proved. Hypothermic Machine Perfusion (HMP) is the mainstream organ perfusion technology. This study aims to compare the effectiveness of NMP with the HMP.

DETAILED DESCRIPTION:
The main purpose of the study is to improve the utilization rate of marginal donors through normothermic perfusion, and reduce the incidence of infection, severe rejection and even graft failure caused by implantation of marginal donors. This study aims at the following aspects:

1. To compare the effects of two methods and perfusion parameters on the quality of marginal donors: normal temperature pulse perfusion and low temperature mechanical perfusion;
2. Explore the methods of evaluating the function of donor organs;
3. Exploring the effects of different mechanical perfusion methods and perfusion conditions on marginal donors;
4. The effect of broad-spectrum antibiotics on improving donor infection through different administration routes and different drug doses during perfusion and preservation.

A single-center prospective randomized controlled study was used to compare the prognosis of renal transplantation between 50 patients with normothermic pulse perfusion and 50 patients with hypothermic mechanical perfusion who were enrolled in our hospital for allograft kidney transplantation.

Assessment factors:

1. Donor parameters: age, sex, creatinine, diabetes, cause of death, length of stay in ICU, calcification of donor renal artery (CRP expression level)
2. Perfusion pressure, perfusion time, perfusion temperature, perfusion vessel resistance index
3. Receptor factors: age, gender, height, weight, BMI, cause of kidney disease (hypertension, diabetes glomerulonephritis, polycystic kidney disease), dialysis time (month), dialysis type (blood/peritoneum), HLA mismatch number, smoking, diabetes, hypertension, heart disease, hyperlipidemia, anemia, complication index (CCI), ASA score (>3 or ≤ 3), operation time, number of donor renal artery branches, number of donor renal vein branches, donor creatinine, cold ischemia time (mins), and the perfusion of the transplanted kidney ( judged by the fluorescence intensity after indocyanine green injection). Laboratory results: PRA (panel-reactive antibody), blood creatinine, estimated glomerular filtration rate (eGFR), blood lactate level, postoperative urine volume. Graft loss, culture result of irrigation solution (bacteria). Sample acquisition: obtaining the blood and urine samples of the recipient and measuring the expression level of globulin A in the serum. In the process of kidney transplantation, the donor's renal artery vessel wall and the recipient's external iliac artery vessel wall were obtained. The blood vessel wall was stained with calcification, CRP to evaluate the calcification of the donor and recipient vessels.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60 years old, gender unlimited
* Volunteer to participate in this clinical trial and sign the informed consent form
* Suffering from end-stage renal disease
* Planned kidney transplantation
* The expanded standard donors (ECD) were obtained

  * The expanded standard kidney donor is defined as: aged cadaver donors over 60 years old or two or three of the following conditions between 50 and 60 years old: death due to cerebrovascular disease; Hypertension; The blood creatinine level before donation was greater than 133umol/L.

Exclusion Criteria:

* Active infection
* Living donor kidney recipient
* Acute rejection
* Second kidney transplantation
* Combined transplantation (combined liver and kidney, combined pancreas and kidney)
* Patients who take other clinical trial drugs or participate in other clinical studies
* Unable to continue the research
* Patients who are judged by the researcher to be unsuitable for this clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-03-03 (Estimated); Primary Completion 2024-12-03 (Estimated); Study Completion 2025-09-03 (Estimated)

PRIMARY OUTCOMES:
Rate of delayed renal function (DGF) | 1 week after surgery
  At least one dialysis is required within one week after kidney transplantation

SECONDARY OUTCOMES:
Estimated glomerular filtration rate | 3, 6, 12 months after surgery
  Calculated from serum creatinine levels to assess kidney function.
Rate of primary non-function (PNF) | 1 months after surgery
  Dialysis is required because the transplanted kidney is nonfunctional
Graft survival and recipient survival | 1 year follow-up
  Incidence of the Graft survival and recipient survival
Complications | within 90 days after operation
  incidence of complications
Patient death | 1 year follow-up
  Death date after surgery and the reasons

OTHER OUTCOMES:
Hospitalization expenses | 3, 6, 12 months after surgery
  Total expenses of kidney transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Zhou Xiaofeng, MD, Study Chair — China-Japan Friendship Hospital
Locations (1):
- China-Japan Friendship Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD, all IPD that underlie results in a publication
Supporting Information: Study Protocol, ICF, CSR
Time Frame: one year after research end
Access Criteria: share the data

REFERENCES:
- [Background] Hamar M, Urbanellis P, Kaths MJ, Kollmann D, Linares I, Ganesh S, Wiebe A, Cen JY, Yip P, John R, Konvalinka A, Mucsi I, Ghanekar A, Bagli D, Grant D, Robinson LA, Selzner M. Normothermic Ex Vivo Kidney Perfusion Reduces Warm Ischemic Injury of Porcine Kidney Grafts Retrieved After Circulatory Death. Transplantation. 2018 Aug;102(8):1262-1270. doi: 10.1097/TP.0000000000002245. PMID 29683999
- [Background] Nicholson ML, Hosgood SA. Renal transplantation after ex vivo normothermic perfusion: the first clinical study. Am J Transplant. 2013 May;13(5):1246-52. doi: 10.1111/ajt.12179. Epub 2013 Feb 22. PMID 23433047
- [Background] Mazilescu LI, Urbanellis P, Kim SJ, Goto T, Noguchi Y, Konvalinka A, Reichman TW, Sayed BA, Mucsi I, Lee JY, Robinson LA, Ghanekar A, Selzner M. Normothermic Ex Vivo Kidney Perfusion for Human Kidney Transplantation: First North American Results. Transplantation. 2022 Sep 1;106(9):1852-1859. doi: 10.1097/TP.0000000000004098. Epub 2022 Mar 1. PMID 35238854
- [Derived] Tingle SJ, Thompson ER, Figueiredo RS, Moir JA, Goodfellow M, Talbot D, Wilson CH. Normothermic and hypothermic machine perfusion preservation versus static cold storage for deceased donor kidney transplantation. Cochrane Database Syst Rev. 2024 Jul 9;7(7):CD011671. doi: 10.1002/14651858.CD011671.pub3. PMID 38979743